CLINICAL TRIAL: NCT04480398
Title: A Retrospective Study on Efficacy and Safety of Guduchi Ghan Vati for Covid-19 Asymptomatic Patients
Brief Title: Efficacy and Safety of Guduchi Ghan Vati for Covid-19 Asymptomatic Patients
Status: Completed | Type: Observational
Sponsor: Aarogyam UK (Other)
Collaborators: Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University (Other); Samta Ayurveda Prakoshtha, India (Unknown)
Responsible Party: Sponsor
Other Study IDs: AYU/DSSR/02
Record Dates: First submitted 2020-07-18; First posted 2020-07-21 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Asymptomatic Condition
Keywords: Ayurveda; Guduchi Ghan Vati
MeSH Terms: conditions — COVID-19; Asymptomatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ayurveda: Guduchi Ghan Vati was given to Covid patients 2 tablets (500 mg each) twice daily were given orally after meal for 28 days. Guduchi ghan vati is a powdered aqueous extract of Tinospora cordifolia in tablet form and prepared in GMP certified Pharmacy of the University, following standard protocol.
  Interventions: Drug: Guduchi Ghan Vati
- Control: Standard care for asymptomatic confirmed cases is isolation (to contain virus transmission) and clinical monitoring as per recommended Guidelines.

INTERVENTIONS:
Drug: Guduchi Ghan Vati — Guduchi Ghan Vati is an Ayuvedic classical preparation which is prepared from aqueous of extract of Tinospora cordifolia.
  Other Names: Giloy Ghan Vati
  Groups: Ayurveda

SUMMARY:
Coronavirus disease 2019 (Covid-19) has been declared global emergency with immediate safety, preventative and curative measures to control the spread of virus. Confirmed cases are treated with clinical management as they are diagnosed but so far, there is no effective treatment or vaccine yet for Covid-19.

With recommended guidelines of AYUSH Ministry, India, the use of Ayurveda for Covid-19 has increased; however, its efficacy and safety in Covid-19 confirmed patients remain unclear.

Present study examined the efficacy and safety of one of the recommended Ayurveda drug (Guduchi Ghan Vati) compared with standard care for patients with asymptomatic Covid-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* A person diagnosed with COVID-19
* Asymptomatic at the time of admission

Exclusion Criteria:

* Patients over 75 years
* Taking antibiotics or antiretroviral for any reason
* Mild to Moderate symptoms at the time of hospital admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Covid-19 Confirmed Asymptomatic patients
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Virologic clearance | 21 days
  Virologic clearance indicates the duration from the first Covid-19 positive result to the first Covid-19 negative result

SECONDARY OUTCOMES:
Change in the number of patients going from asymptomatic to moderately disease | 10-days of hospital admission
  change in the number of patients going from asymptomatic to moderately disease
Hospital Stay | 21 days
  Total duration of stay in hospital for complete recovery
Clinically relevant adverse effects | 21-days
  Clinically relevant adverse effects of Guduchi Ghan Vati (Disability, Discomfort reported)

CONTACTS AND LOCATIONS:
Overall Officials: Parashar Sharma, Study Chair — Samta Ayurveda Prakoshtha; Jaydeep Joshi, Study Chair — Aarogyam UK; Neha Sharma, Study Director — Aarogyam UK; Abhimanyu Kumar, Principal Investigator — Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University
Locations (1):
- Dr Sarvepalli Radhakrishnan Rajasthan Ayurved University, Jodhpur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided